CLINICAL TRIAL: NCT01321255
Title: Improving Equitable Acces and Adherence to Secondary Prevention Therapy With a Fixed-Dose Combination Drug
Brief Title: Fixed Dose Combination Drug (Polypill)for Secondary Cardiovascular Prevention.
Acronym: FOCUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Centro Nacional de Investigaciones Cardiovasculares Carlos III (Other)
Collaborators: Mario Negri Institute for Pharmacological Research (Other); Rusculleda Foundation Instituto DAMIC (Unknown); Fundacion Clinic per a la Recerca Biomédica (Other); ARTTIC International Management Services (Unknown); Federación Argentina de Cardiología FAC (Unknown); World Health Organization (Other); Instituto de Salud Carlos III (Other Government); Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FOCUS; 2010-022492-54 (EudraCT Number); Health-F2-2009-241559 (Other Grant/Funding Number: Frame of Seventh Investigation Marco Programme, Technological development and Innovation of the EU)
Record Dates: First submitted 2011-03-21; First posted 2011-03-23 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Treatment Adherence
MeSH Terms: conditions — Myocardial Infarction; Treatment Adherence and Compliance | interventions — Simvastatin; Aspirin; Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FDC Fixed Dose Combination (Experimental)
  Interventions: Drug: FDC
- Conventional treatment (Active Comparator)
  Interventions: Drug: Separately drugs, simvastatin, aspirin and ramipril

INTERVENTIONS:
Drug: FDC — FDC includes a combination of 100 mg aspirin, 40 mg simvastatin, and 2.5;5;10 mg Ramipril
  Arms: FDC Fixed Dose Combination
Drug: Separately drugs, simvastatin, aspirin and ramipril — Aspirin 100 mg once a day Ramipril 2.5; 5; 10 mg once a day Simvastatin 40 mg once a day
  Arms: Conventional treatment

SUMMARY:
The aim of the FOCUS project is to test the Fixed Dose Combination concept for cardiovascular prevention in populations of different socio-economic characteristics. At the same time, FOCUS aims to understand the factors determining inappropriate prescribing for secondary cardiovascular prevention and those for poor patients adherence to treatment. This will allow FOCUS to establish recommendations for a better use of medication in patients with ischemic heart disease. In addition, after a successful completion of FOCUS, secondary prevention medication will be available and affordable for a large number of patients in both developed as well as developing countries.

There are two Phases in this study:

Phase 1: Is a descriptive, non interventional study. Phase 2: Is an interventional, randomized trial with prospective economic evaluation.

DETAILED DESCRIPTION:
The specific objective of the FOCUS project is to prove that:

1. Better knowledge of factors relates to inappropriate use of secondary cardiovascular prevention drugs and lack of adherence to treatment will help to design new strategies for improving patients' management.
2. A Fixed Dose Combination (FDC, polypill) including three components with a well demonstrated efficacy will improve secondary prevention in coronary patients by decreasing inappropriate prescribing and by reducing complexity of treatment and lack of adherence.

   * Phase 1 is a descriptive, non-interventional study. Its aim is to provide a comprehensive analysis of potential factors precluding adequate secondary prevention, including Health system characteristics, drugs affordability and availability, as well as patients' characteristics. Differences between the two studied regions (Europe and South America) will be analyzed.
   * Phase 2 is an interventional, randomized trial with prospective economic evaluation. It will be organised as a two-arm, randomised, parallel, multinational study. Patients completing the Phase 1, and fulfilling inclusion/exclusion criteria (see below), will be included in Phase 2. Patients will be randomized to receive a FDC of ramipril, simvastatin and acetylsalicylic acid or the three medications separately.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1: All patients, male and female, 40 years of age or older, with a history of ST-elevation AMI within the last 2 years, attending any of the selected sites and signing the consent
* Phase 2: All patients, male and female, 40 years of age or older, with a history of ST-elevation AMI within the last 2 years, attending any of the selected sites and signing the consent Patients in whom secondary prevention with ASA, statin and ACEI is indicated, Signing informed consent

Exclusion Criteria:

* Phase 1: Patients in which any of the components of the FDC is contraindicated. Living in a nursing home. Memtal illness limiting the capacity of
* Phase 2:Secondary dyslipemia, Patients in which any of the components of the FDC is contraindicated, Living in a nursing home, Mental illness limiting the capacity of self care, Participating in another trial, , Previous Percutaneous Transluminal Coronary Angioplasty (PTCA) with a drug eluting stent (DES) whitin the last year, Severe Congestive Heart Failure (NYHA III-IV), Serum creatinine >2 mg/dl, any condition limiting life expectancy <2 years. Pregnant or premenopausal women.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2118 (Actual)
Dates: Start 2012-01; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients receiving AAS, an ACE inhibitor and a statin among those without contraindications to any of these drugs Adherence to treatment measured by: Morinsky-Green test and Pill accountability. | 18 months
  Phase 1
Adherence to treatment measured by the Morisky-Green questionnaire | 18 months
  Phase 1:
  Adherence to treatment measured by the Morisky-Green questionnaire. According to this, patients will be classified as "Good adherents" when the total score ranges between 16 and 20 and as "Poor adherents" if the total score is <16 points
Treatment adherence measured by: Morisky-Green test: (Good adherence score 16-20) at 1 and 9 months. | 18 months
  Phase 2
Treatment adherence measured by: Pill counts at 1-4-9 months. (Good adherence 80-110% PC) | 18 months
  Phase 2

SECONDARY OUTCOMES:
Blood Pressure and Lipid Profile (LDL-cholesterol) at 1 and 9 months | 18 months
  Phase 2
Safety and tolerability: Adverse events and rate of treatment withdrawal. | 18 months
  Phase 2

CONTACTS AND LOCATIONS:
Overall Officials: Valentín Fuster, MD PhD, Principal Investigator — Centro Nacional de Investigaciones Cardiovasculares Carlos III; Ginés Sanz, MD PhD, Study Director — Centro Nacional de Investigaciones Cardiovasculares Carlos III
Locations (69):
- Argentina (25):
  - Sanatorio Güemes, Buenos Aires
  - CENUDIAB, Buenos Aires
  - Centro Médico GEA 3 Privado, Córdoba
  - Hospital San Roque, Córdoba
  - Hospital Nuestra Señora de la Misericordia, Córdoba
  - Clínica Colombo, Córdoba
  - Instituto Médico DAMIC, Córdoba
  - Hospital Italiano, Córdoba
  - Hospital de Córdoba, Córdoba
  - Sanatorio Parque S.A., Córdoba
  - IPAC - Clínica Privada Caraffa S.R.L., Córdoba
  - Consultan Salud S.A., Haedo
  - Hospital Italiano, La Plata
  - Fundación CICLO, La Plata
  - Clínica Constituyentes, Morón
  - Instituto de Investigaciones Clínicas Quilmes, Quilmes
  - DIM Clínica Privada, Ramos Mejía
  - Sanatorio Británico S.A., Rosario
  - Hospital Italiano de Rosario Garibaldi, Rosario
  - Hospital Provincial del Centenario, Rosario
  - Sanatorio Julio Corzo, Rosario
  - Corporación Médica General San Martín, San Martín
  - Clínica Privada de la Ciudad S.R.L., Villa Allende
  - Sanatorio Cruz Azul S.R.L., Villa María
  - Clínica Privada de Especialidades de Villa María S.R.L., Villa María
- Brazil (5):
  - INOVAR Pesquisas clínicas, São Paulo
  - Centro de Pesquisa SeÇão de Hipeertensão e Nefrología - Instituto Dante Pazzanese, São Paulo
  - Nefrología Centro de Pesquisa Clínica do Hospital do Rim e Hipertensão, São Paulo
  - UNIFESP - Setor de Lípides, Atersclerose e Biologia Vascular, São Paulo
  - Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
- Italy (14):
  - Ospedale F. Ferrari, Casarano
  - Azienda Istituti Ospitalieri, Cremona
  - Presidio Ospedaliero di Desio, Desio
  - Ospedale S. Cuore di Gesù, Gallipoli
  - Ospedale F. Veneziale, Isernia
  - Ospedale Niguarda Cá Granda, Milan
  - Azienda Ospedaler San Gerardo, Monza
  - Ospedale Civile San Francesco di Paola, Paola
  - Azienda Ospedale G. Salvani - Presidio di Passirana, Passirana Di Rho
  - Ospedale Fondazione Salvatore Maugeri, Pavia
  - Ospedale Sant´ Antonio, San Daniele
  - Ospedale San Bartolomeo, Sarzana
  - Presidio Ospedaliero di Sondrio, Sondrio
  - Casa di Cura - Villa Bianca, Trento
- Paraguay (4):
  - Hospital Central del Instituto de Previsión Social (HC-IPS), Asunción
  - Hospital Universitario Nuestra Señora de la Asunción, Asunción
  - Hospitalñ de Clínicas - Catedra de Semiologia Médica - Universidad Nacional de Asunción, Asunción
  - Hospital Nacional de Itagua, Itauguá
- Spain (21):
  - Hospital Principes de Asturias, Alcalá de Henares, Madrid
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - CS Aldaia, Aldaia, Valencia
  - CS Cheste, Cheste, Valencia
  - CS Manises, Manises, Valencia
  - CS Ribarroja del Túria, Ribarroja del Turia, Valencia
  - Hospital General de Alicante, Alicante
  - EAP Poble Sec, Barcelona
  - CAP Vallcarca, Barcelona
  - ABS Gaudi, Barcelona
  - EAP Sardenya, Barcelona
  - Hospital Sant Pau, Barcelona
  - EAP Sarrià, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital La Princesa, Madrid
  - CS Ángela Uriarte, Madrid
  - CS San Andrés III, Madrid
  - CS Villablanca, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Virgen Arrixaca, Murcia
  - Hospital Virgen Macarena, Seville

REFERENCES:
- [Background] World Health Organization. Price, availability and affordability. An international comparison of chronic disease medicines. Background report prepared for the WHO Plannig Meeting on the Global Initiative for Treatment of Chronic Diseases, Cairo, December 2005
- [Background] European Cardiovascular Disease Statistics. British Heart Foundation and European Heart Network. 2005
- [Background] European Health Heart Charter. Available at www.heartcharter.eu
- [Background] Beaglehole R, Reddy S, Leeder SR. Poverty and human development: the global implications of cardiovascular disease. Circulation. 2007 Oct 23;116(17):1871-3. doi: 10.1161/CIRCULATIONAHA.107.736926. No abstract available. PMID 17965400
- [Background] kaplan W. LR. Priority medicines for Europe and the World; 2004 November.
- [Background] Reddy KS. Cardiovascular diseases in the developing countries: dimensions, determinants, dynamics and directions for public health action. Public Health Nutr. 2002 Feb;5(1A):231-7. doi: 10.1079/phn2001298. PMID 12027289
- [Background] Ezzati M, Lopez AD. Estimates of global mortality attributable to smoking in 2000. Lancet. 2003 Sep 13;362(9387):847-52. doi: 10.1016/S0140-6736(03)14338-3. PMID 13678970
- [Background] Mackenbach JP, Stirbu I, Roskam AJ, Schaap MM, Menvielle G, Leinsalu M, Kunst AE; European Union Working Group on Socioeconomic Inequalities in Health. Socioeconomic inequalities in health in 22 European countries. N Engl J Med. 2008 Jun 5;358(23):2468-81. doi: 10.1056/NEJMsa0707519. PMID 18525043
- [Background] Asaria P, Chisholm D, Mathers C, Ezzati M, Beaglehole R. Chronic disease prevention: health effects and financial costs of strategies to reduce salt intake and control tobacco use. Lancet. 2007 Dec 15;370(9604):2044-53. doi: 10.1016/S0140-6736(07)61698-5. Epub 2007 Dec 11. PMID 18063027
- [Background] Yusuf S, Hawken S, Ounpuu S, Dans T, Avezum A, Lanas F, McQueen M, Budaj A, Pais P, Varigos J, Lisheng L; INTERHEART Study Investigators. Effect of potentially modifiable risk factors associated with myocardial infarction in 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):937-52. doi: 10.1016/S0140-6736(04)17018-9. PMID 15364185
- [Background] Lopez AD, Mathers CD, Ezzati M, Jamison DT, Murray CJ. Global and regional burden of disease and risk factors, 2001: systematic analysis of population health data. Lancet. 2006 May 27;367(9524):1747-57. doi: 10.1016/S0140-6736(06)68770-9. PMID 16731270
- [Background] Sanz GA. [Risk stratification in acute coronary syndromes: an unresolved issue]. Rev Esp Cardiol. 2007 Oct;60 Suppl 3:23-30. Spanish. PMID 18093491
- [Background] Granger CB, Goldberg RJ, Dabbous O, Pieper KS, Eagle KA, Cannon CP, Van De Werf F, Avezum A, Goodman SG, Flather MD, Fox KA; Global Registry of Acute Coronary Events Investigators. Predictors of hospital mortality in the global registry of acute coronary events. Arch Intern Med. 2003 Oct 27;163(19):2345-53. doi: 10.1001/archinte.163.19.2345. PMID 14581255
- [Background] Chiuve SE, McCullough ML, Sacks FM, Rimm EB. Healthy lifestyle factors in the primary prevention of coronary heart disease among men: benefits among users and nonusers of lipid-lowering and antihypertensive medications. Circulation. 2006 Jul 11;114(2):160-7. doi: 10.1161/CIRCULATIONAHA.106.621417. Epub 2006 Jul 3. PMID 16818808
- [Background] Davies AR, Smeeth L, Grundy EM. Contribution of changes in incidence and mortality to trends in the prevalence of coronary heart disease in the UK: 1996 2005. Eur Heart J. 2007 Sep;28(17):2142-7. doi: 10.1093/eurheartj/ehm272. Epub 2007 Jul 18. PMID 17636307
- [Background] Antithrombotic Trialists' Collaboration. Collaborative meta-analysis of randomised trials of antiplatelet therapy for prevention of death, myocardial infarction, and stroke in high risk patients. BMJ. 2002 Jan 12;324(7329):71-86. doi: 10.1136/bmj.324.7329.71. PMID 11786451
- [Background] Baigent C, Keech A, Kearney PM, Blackwell L, Buck G, Pollicino C, Kirby A, Sourjina T, Peto R, Collins R, Simes R; Cholesterol Treatment Trialists' (CTT) Collaborators. Efficacy and safety of cholesterol-lowering treatment: prospective meta-analysis of data from 90,056 participants in 14 randomised trials of statins. Lancet. 2005 Oct 8;366(9493):1267-78. doi: 10.1016/S0140-6736(05)67394-1. Epub 2005 Sep 27. PMID 16214597
- [Background] Smith SC Jr, Allen J, Blair SN, Bonow RO, Brass LM, Fonarow GC, Grundy SM, Hiratzka L, Jones D, Krumholz HM, Mosca L, Pasternak RC, Pearson T, Pfeffer MA, Taubert KA; AHA/ACC; National Heart, Lung, and Blood Institute. AHA/ACC guidelines for secondary prevention for patients with coronary and other atherosclerotic vascular disease: 2006 update: endorsed by the National Heart, Lung, and Blood Institute. Circulation. 2006 May 16;113(19):2363-72. doi: 10.1161/CIRCULATIONAHA.106.174516. No abstract available. PMID 16702489
- [Background] Fletcher GF, Bufalino V, Costa F, Goldstein LB, Jones D, Smaha L, Smith SC Jr, Stone N. Efficacy of drug therapy in the secondary prevention of cardiovascular disease and stroke. Am J Cardiol. 2007 Mar 27;99(6C):1E-35E. doi: 10.1016/j.amjcard.2007.02.001. Epub 2007 Mar 5. No abstract available. PMID 17378996
- [Background] Dagenais GR, Pogue J, Fox K, Simoons ML, Yusuf S. Angiotensin-converting-enzyme inhibitors in stable vascular disease without left ventricular systolic dysfunction or heart failure: a combined analysis of three trials. Lancet. 2006 Aug 12;368(9535):581-8. doi: 10.1016/S0140-6736(06)69201-5. PMID 16905022
- [Background] Danchin N, Cucherat M, Thuillez C, Durand E, Kadri Z, Steg PG. Angiotensin-converting enzyme inhibitors in patients with coronary artery disease and absence of heart failure or left ventricular systolic dysfunction: an overview of long-term randomized controlled trials. Arch Intern Med. 2006 Apr 10;166(7):787-96. doi: 10.1001/archinte.166.7.787. PMID 16606817
- [Background] Doval HCT, C.D. Prevención secundaria de las enfermedades cardiovasculares. In: Evidencias en Cardiología. Buenos Aires: GEDIC; 2008.
- [Background] Law MR, Wald NJ, Rudnicka AR. Quantifying effect of statins on low density lipoprotein cholesterol, ischaemic heart disease, and stroke: systematic review and meta-analysis. BMJ. 2003 Jun 28;326(7404):1423. doi: 10.1136/bmj.326.7404.1423. PMID 12829554
- [Background] Mendis S, Abegunde D, Yusuf S, Ebrahim S, Shaper G, Ghannem H, Shengelia B. WHO study on Prevention of REcurrences of Myocardial Infarction and StrokE (WHO-PREMISE). Bull World Health Organ. 2005 Nov;83(11):820-9. Epub 2005 Nov 10. PMID 16302038
- [Background] Antithrombotic Trialists' (ATT) Collaboration; Baigent C, Blackwell L, Collins R, Emberson J, Godwin J, Peto R, Buring J, Hennekens C, Kearney P, Meade T, Patrono C, Roncaglioni MC, Zanchetti A. Aspirin in the primary and secondary prevention of vascular disease: collaborative meta-analysis of individual participant data from randomised trials. Lancet. 2009 May 30;373(9678):1849-60. doi: 10.1016/S0140-6736(09)60503-1. PMID 19482214
- [Background] EUROASPIRE I and II Group; European Action on Secondary Prevention by Intervention to Reduce Events. Clinical reality of coronary prevention guidelines: a comparison of EUROASPIRE I and II in nine countries. EUROASPIRE I and II Group. European Action on Secondary Prevention by Intervention to Reduce Events. Lancet. 2001 Mar 31;357(9261):995-1001. doi: 10.1016/s0140-6736(00)04235-5. PMID 11293642
- [Background] Heras M, Marrugat J, Aros F, Bosch X, Enero J, Suarez MA, Pabon P, Ancillo P, Loma-Osorio A, Rodriguez JJ, Subirana I, Vila J; en representacion de los investigadores del estudio PRIAMHO. [Reduction in acute myocardial infarction mortality over a five-year period]. Rev Esp Cardiol. 2006 Mar;59(3):200-8. Spanish. PMID 16712743
- [Background] Kotseva K. Global preventive policies. Strategies at European and worldwide level. Rev Esp Cardiol. 2008 Sep;61(9):960-70. English, Spanish. PMID 18775238
- [Background] Kristensen SD, Baumgartner H, Drexler H, Eeckhout E, Filippatos G, Gitt AK, Linde C, Pierard LA, Poldermans D, Schunkert H, Sipido KR, van der Wall EE, Fox K, Bax JJ; European Society of Cardiology. Highlights of the 2007 scientific sessions of the European Society of Cardiology Vienna, Austria, September 1-5, 2007. J Am Coll Cardiol. 2007 Dec 18;50(25):2421-30. doi: 10.1016/j.jacc.2007.10.010. No abstract available. PMID 18154969
- [Background] Mendis S, Fukino K, Cameron A, Laing R, Filipe A Jr, Khatib O, Leowski J, Ewen M. The availability and affordability of selected essential medicines for chronic diseases in six low- and middle-income countries. Bull World Health Organ. 2007 Apr;85(4):279-88. doi: 10.2471/blt.06.033647. PMID 17546309
- [Background] Trust WW. Second World Health Organization & Wellcome Trust Workshop. In: Secondary Prevention of Cardiovascular Disease in Low & Middle Income Countries - Building the Evidence Base on Secondary Prevention of CVD. 2007 6-8 June; London; 2007
- [Background] Kotseva K, Wood D, De Backer G, De Bacquer D, Pyorala K, Keil U; EUROASPIRE Study Group. Cardiovascular prevention guidelines in daily practice: a comparison of EUROASPIRE I, II, and III surveys in eight European countries. Lancet. 2009 Mar 14;373(9667):929-40. doi: 10.1016/S0140-6736(09)60330-5. PMID 19286092
- [Background] Gaziano TA, Galea G, Reddy KS. Scaling up interventions for chronic disease prevention: the evidence. Lancet. 2007 Dec 8;370(9603):1939-46. doi: 10.1016/S0140-6736(07)61697-3. PMID 18063028
- [Background] Gaziano TA. Economic burden and the cost-effectiveness of treatment of cardiovascular diseases in Africa. Heart. 2008 Feb;94(2):140-4. doi: 10.1136/hrt.2007.128785. PMID 18195120
- [Background] Beaglehole R, Ebrahim S, Reddy S, Voute J, Leeder S; Chronic Disease Action Group. Prevention of chronic diseases: a call to action. Lancet. 2007 Dec 22;370(9605):2152-7. doi: 10.1016/S0140-6736(07)61700-0. Epub 2007 Dec 11. PMID 18063026
- [Background] Pharma 2020: the vision. Which path will you take? (Accessed at http://www.pwc.com/pharma.)
- [Background] Bosworth HB. Medication treatment adherence. Chapter 6, 147-94. In: Bosworth H, Oddone, E., Weinberger, M., ed. In:
- [Background] DiMatteo MR. Variations in patients' adherence to medical recommendations: a quantitative review of 50 years of research. Med Care. 2004 Mar;42(3):200-9. doi: 10.1097/01.mlr.0000114908.90348.f9. PMID 15076819
- [Background] Gehi A, Haas D, Pipkin S, Whooley MA. Depression and medication adherence in outpatients with coronary heart disease: findings from the Heart and Soul Study. Arch Intern Med. 2005 Nov 28;165(21):2508-13. doi: 10.1001/archinte.165.21.2508. PMID 16314548
- [Background] DiMatteo MR, Lepper HS, Croghan TW. Depression is a risk factor for noncompliance with medical treatment: meta-analysis of the effects of anxiety and depression on patient adherence. Arch Intern Med. 2000 Jul 24;160(14):2101-7. doi: 10.1001/archinte.160.14.2101. PMID 10904452
- [Background] DiMatteo MR. Social support and patient adherence to medical treatment: a meta-analysis. Health Psychol. 2004 Mar;23(2):207-18. doi: 10.1037/0278-6133.23.2.207. PMID 15008666
- [Background] Rasmussen JN, Chong A, Alter DA. Relationship between adherence to evidence-based pharmacotherapy and long-term mortality after acute myocardial infarction. JAMA. 2007 Jan 10;297(2):177-86. doi: 10.1001/jama.297.2.177. PMID 17213401
- [Background] Mukherjee D, Fang J, Chetcuti S, Moscucci M, Kline-Rogers E, Eagle KA. Impact of combination evidence-based medical therapy on mortality in patients with acute coronary syndromes. Circulation. 2004 Feb 17;109(6):745-9. doi: 10.1161/01.CIR.0000112577.69066.CB. PMID 14970110
- [Background] Ho PM, Spertus JA, Masoudi FA, Reid KJ, Peterson ED, Magid DJ, Krumholz HM, Rumsfeld JS. Impact of medication therapy discontinuation on mortality after myocardial infarction. Arch Intern Med. 2006 Sep 25;166(17):1842-7. doi: 10.1001/archinte.166.17.1842. PMID 17000940
- [Background] Danchin N, Cambou JP, Hanania G, Kadri Z, Genes N, Lablanche JM, Blanchard D, Vaur L, Clerson P, Gueret P; USIC 2000 investigators. Impact of combined secondary prevention therapy after myocardial infarction: data from a nationwide French registry. Am Heart J. 2005 Dec;150(6):1147-53. doi: 10.1016/j.ahj.2005.01.058. PMID 16338251
- [Background] Jackevicius CA, Li P, Tu JV. Prevalence, predictors, and outcomes of primary nonadherence after acute myocardial infarction. Circulation. 2008 Feb 26;117(8):1028-36. doi: 10.1161/CIRCULATIONAHA.107.706820. PMID 18299512
- [Background] World Bank Report: Public Policy and the Challenge of Chronic Noncommunicable Diseases. 2007. (Accessed at http://siteresources.worldbank.org/INTPH/Resources/PublicPolicyandNCDsWorldBank2007FullReport.pdf.)
- [Background] Wald NJ, Law MR. A strategy to reduce cardiovascular disease by more than 80%. BMJ. 2003 Jun 28;326(7404):1419. doi: 10.1136/bmj.326.7404.1419. PMID 12829553
- [Background] Wise J. Polypill holds promise for people with chronic disease. Bull World Health Organ. 2005 Dec;83(12):885-7. Epub 2006 Jan 30. No abstract available. PMID 16462975
- [Background] Sleight P, Pouleur H, Zannad F. Benefits, challenges, and registerability of the polypill. Eur Heart J. 2006 Jul;27(14):1651-6. doi: 10.1093/eurheartj/ehi841. Epub 2006 Apr 7. PMID 16603580
- [Background] Reddy KS. Is a multidrug regimen cost-effective for the prevention of cardiovascular disease in resource-poor countries? Nat Clin Pract Cardiovasc Med. 2007 Mar;4(3):130-2. doi: 10.1038/ncpcardio0799. Epub 2007 Jan 30. No abstract available. PMID 17262058
- [Background] Reddy KS. The preventive polypill--much promise, insufficient evidence. N Engl J Med. 2007 Jan 18;356(3):212. doi: 10.1056/NEJMp068219. No abstract available. PMID 17229947
- [Background] Herrick TM, Million RP. Tapping the potential of fixed-dose combinations. Nat Rev Drug Discov. 2007 Jul;6(7):513-4. doi: 10.1038/nrd2334. No abstract available. PMID 17715499
- [Background] Fuster V, Sanz G. A polypill for secondary prevention: time to move from intellectual debate to action. Nat Clin Pract Cardiovasc Med. 2007 Apr;4(4):173. doi: 10.1038/ncpcardio0858. No abstract available. PMID 17380163
- [Background] Combination Pharmacotherapy and Public Health Research Working Group. Combination pharmacotherapy for cardiovascular disease. Ann Intern Med. 2005 Oct 18;143(8):593-9. doi: 10.7326/0003-4819-143-8-200510180-00010. PMID 16230726
- [Background] Bangalore S, Kamalakkannan G, Parkar S, Messerli FH. Fixed-dose combinations improve medication compliance: a meta-analysis. Am J Med. 2007 Aug;120(8):713-9. doi: 10.1016/j.amjmed.2006.08.033. PMID 17679131
- [Background] Dickson M, Plauschinat CA. Compliance with antihypertensive therapy in the elderly: a comparison of fixed-dose combination amlodipine/benazepril versus component-based free-combination therapy. Am J Cardiovasc Drugs. 2008;8(1):45-50. doi: 10.2165/00129784-200808010-00006. PMID 18303937
- [Background] Pan F, Chernew ME, Fendrick AM. Impact of fixed-dose combination drugs on adherence to prescription medications. J Gen Intern Med. 2008 May;23(5):611-4. doi: 10.1007/s11606-008-0544-x. Epub 2008 Feb 21. PMID 18288541
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Radloff LS. The CES-D scale: a self-report depression scale for research in the general population. Applied Psychology Measurements 1977;1.
- [Background] Berkman LF, Blumenthal J, Burg M, Carney RM, Catellier D, Cowan MJ, Czajkowski SM, DeBusk R, Hosking J, Jaffe A, Kaufmann PG, Mitchell P, Norman J, Powell LH, Raczynski JM, Schneiderman N; Enhancing Recovery in Coronary Heart Disease Patients Investigators (ENRICHD). Effects of treating depression and low perceived social support on clinical events after myocardial infarction: the Enhancing Recovery in Coronary Heart Disease Patients (ENRICHD) Randomized Trial. JAMA. 2003 Jun 18;289(23):3106-16. doi: 10.1001/jama.289.23.3106. PMID 12813116
- [Derived] Castellano JM, Sanz G, Penalvo JL, Bansilal S, Fernandez-Ortiz A, Alvarez L, Guzman L, Linares JC, Garcia F, D'Aniello F, Arnaiz JA, Varea S, Martinez F, Lorenzatti A, Imaz I, Sanchez-Gomez LM, Roncaglioni MC, Baviera M, Smith SC Jr, Taubert K, Pocock S, Brotons C, Farkouh ME, Fuster V. A polypill strategy to improve adherence: results from the FOCUS project. J Am Coll Cardiol. 2014 Nov 18-25;64(20):2071-82. doi: 10.1016/j.jacc.2014.08.021. Epub 2014 Sep 1. PMID 25193393
- [Derived] Sanz G, Fuster V, Guzman L, Guglietta A, Arnaiz JA, Martinez F, Sarria A, Roncaglioni MC, Taubert K. The fixed-dose combination drug for secondary cardiovascular prevention project: improving equitable access and adherence to secondary cardiovascular prevention with a fixed-dose combination drug. Study design and objectives. Am Heart J. 2011 Nov;162(5):811-817.e1. doi: 10.1016/j.ahj.2011.08.012. PMID 22093195
- See also: CNIC — http://www.cnic.es/en/index.php